CLINICAL TRIAL: NCT03278990
Title: A Test of Scalable Behavioral Interventions to Increase PrEP Adherence for At-Risk HIV- Individuals: Value Affirmation and Future Selves
Brief Title: Scalable Interventions to Increase PrEP Adherence: Value Affirmation and Future Selves
Acronym: SIIPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not meet recruitment goals
Sponsor: Stuart Fisk (Other)
Collaborators: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); Gilead Sciences (Industry); University of Pittsburgh (Other); Allies for Health + Wellbeing (Unknown); Center for Inclusion Health, Allegheny General Hospital (Unknown); Metro Community Health Center (Unknown)
Responsible Party: Sponsor-Investigator, Stuart Fisk, Sponsor-Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IN-US-276-4221
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: HIV Prevention
Keywords: PrEP; Prevention; Value Affirmation; Future Selves; Behavioral Intervention

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized trial with 2 arms-a control arm with allocation ratio of 50%, and an intervention arm (future self-value affirmation) with an allocation ratio of 50%.
Who Masked: Participant, Care Provider
Masking Description: Participants are randomly assigned to treatment or control exercises involving writing for 5 minutes. Participants do not know there is another writing condition. Care providers do not see the written content provided by the participant. Neither the participants nor the care provider will know which condition the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Future Self - Value Affirmation (Experimental): This is a behavioral intervention whereby participants write (Value Affirmation and Future Selves Combination) for 5 minutes about 1-2 values that are important to them, as well as about a time in their life when they were particularly important. Next, for five minutes, they write a letter to themselves in 20 years.
  Interventions: Behavioral: Value Affirmation and Future Selves Combination
- Control (Sham Comparator): In this sham comparator, participants will also write (Control Writing Exercise) --similar to the intervention above. However, the content of the writing exercise is different. Participants write for five minutes about what they did that day. Next, for five minutes, they write a letter to themselves next week.
  Interventions: Behavioral: Control writing exercise

INTERVENTIONS:
Behavioral: Value Affirmation and Future Selves Combination — Following the questionnaire, participants will complete a 10- to 15-minute writing exercise. In the control condition, they will be given a list of values, select two that are least important to them, then write about why those values might be important to others. Next, they will write a short letter to themselves in 2 weeks. In the treatment condition, they will be given a list of values, select two that are important to them, then write for about why those values are important to them and how they have played a role in their life. They will then write a short letter to themselves twenty years in the future.
  Arms: Future Self - Value Affirmation
Behavioral: Control writing exercise — In this sham comparator, participants will also write, however, the content of the writing exercise is different. Participants write for five minutes about what they did that day. Next, for five minutes, they write a letter to themselves next week.
  Arms: Control

SUMMARY:
Pre-exposure prophylaxis, or PrEP, is a relatively new HIV prevention method where individuals who are at risk for HIV but do not currently have it take a daily pill (Truvada). PrEP has been proven medically effective and could help to reduce the rate of new HIV incidence in the United States, but in five large, randomized and controlled studies, many prospective PrEP patients chose not to take PrEP, and those that did often did not adhere to it consistently. How do we increase PrEP uptake and adherence amongst those most at risk for HIV? Also, will taking PrEP increase or decrease high-risk individual sexual behavior and HIV incidence? Here, the investigators propose a parallel group randomized, controlled clinical trial to test the effectiveness of a behavioral intervention designed to buffer individuals against stigma-related feelings, and to increase their connection to their selves twenty years in the future. The primary objective of the study is to increase PrEP adherence, as measured by the concentration of tenofovir diphosphate (TFV-DP) in dried blood spot samples (DBS). The secondary objectives are to decrease the incidence of STIs and increase safe sexual practices, as measured by clinic diagnoses and self-reported practices at 3, 6, 9 and 12 months.

This 12-month outpatient study will take place at four PrEP clinics in Pittsburgh and will enroll 170 subjects across 4 sites, with an expectation of retaining 80%, or 135 subjects. Eligibility includes male and female adults, ages 18-65, who are at risk of contracting HIV. Efforts will be made to recruit 33% of subjects from each of the following strata: 1) young, minority LGBT adults age 18-30 years of age; 2) Caucasian adults (MSM and heterosexual females) age 18-65 years of age; and 3) IDU adults, age 18-65, of any ethnic background.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis, or PrEP, is a relatively new HIV prevention method where individuals who are at risk for HIV but do not currently have it take a daily pill (Truvada). The CDC currently recommends PrEP as a method of HIV prevention in high-risk individuals based on compelling efficacy data from large international studies in diverse populations, but the issue of adherence and its relationship to clinical efficacy is still being defined. In five large, randomized and controlled studies, many prospective PrEP patients chose not to take PrEP, and those that did often did not adhere to it consistently (Landovitz & Coates, 2014). Experts remain unable to answer several high-stakes questions: How do we increase PrEP uptake and adherence amongst those most at risk for HIV, and will starting PrEP increase or decrease high-risk individual sexual behavior and HIV incidence? (Landovitz & Coates, 2014). In sum, the biggest challenge to reducing new HIV incidence in the U.S. is behavioral, not medical.

Here, the investigators propose a randomized, controlled clinical study to test the effectiveness of a "future selves-value affirmation" behavioral intervention on PrEP uptake and adherence. The intervention is designed to address the challenges of stigma and "present bias" - the individual propensity to place the gains of the moment ahead of future gains- as it relates to adherence.

"Present bias" and the suboptimal decisions it produces derive from a limited ability to imagine one's self in the future, and lead to a patient's preference for smaller, immediate rewards (e.g., escaping side effects of a medication, safeguarding one's situation from loved ones) over larger, delayed ones (e.g., not contracting HIV, longer life expectancy, better health). Research has shown that vivid, concrete, and detailed images of one's future self enhance a person's ability to envision and emotionally engage the future consequences of present-day decisions. For instance, creating positive images of one's future self has been shown to stem delinquent behavior for up to a year (van Gelder, 2013).

To address stigma, the investigators draw on another literature in psychology which has now established that short value affirmation exercises are able to enhance learning, performance, control and commitment outcomes, and to do so most effectively with populations facing stigma in the domain of interest (Vohs & Smeichel, 2009; Creswell et al., 2013; Creswell & Lindsay, 2014), especially within the domain of health behavior change (Ehret & Sherman, 2014; Harris, 2011; Reed & Aspinwall, 1998; Nustad, 2011; Cohen and Sherman, 2014; Epton et al., 2015). Affirmation exercises can be as simple as writing or talking for 5 minutes about a value one holds dear. Indeed, one such 5-minute exercise at the beginning of a new program or project can lead to profoundly powerful long-term outcomes across very different settings. For example, one intervention led to a .41 point grade increase for minority students in college over the course of one and two years (Cohen et al, 2009), increased decision making skills and use of public service information by homeless shelter participants in Seattle (Hall et al., 2014), and enabled smokers to more readily accept threatening smoking risk information (Epton et al., 2015). This study will combine value affirmation and future selves approaches.

The first study objective is to evaluate the effect of the "future-selves / value affirmation" intervention on PrEP adherence, as measured by tenofovir levels in dried blood spots and categorized via the 5-level ordinal measure for Engagement with PrEP (used in the iPrEx Open-Label Extension). The secondary study objectives are to evaluate the effect of the "future-selves / value affirmation" intervention on HIV and STI contraction at 3, 6, 9, and 12 months, and to evaluate the effect of the "future-selves / value affirmation" intervention on sexual risk behaviors, as self-reported numbers of anal/vaginal sex partners and episodes of condomless receptive anal and vaginal sex at 3, 6, 9 and 12 months.

This is a parallel group randomized trial with 2 arms-a control arm with allocation ratio of 50%, and an intervention arm (future self-value affirmation) with an allocation ratio of 50%. At each clinic visit, participants will engage in a 10-minute writing (or oral, for those with literacy challenges) exercises. Participants in the intervention arm will be given a list of values, asked to select one that has been particularly important to them at critical times in their life, then asked to write about why that value is important to them. Next, those same participants will write a letter to themselves twenty (20) years in the future. Participants in the control arm will first write for 5 minutes about why two values that are least important to them may be important to someone else, and next write a letter to themselves two weeks in the future.

The study includes 170 subjects enrolled across 4 sites in Pittsburgh, with an expectation of retaining 80%, or 135 subjects. Each subject's participation will last for 12 months.The entire study is expected to last for 18 months. The investigators will evaluate concentrations of tenofovir diphosphate (TFV-DP) in dried blood spot samples at baseline and then quarterly visits; they will also perform quarterly evaluations of self-reported numbers of anal/vaginal sex partners and episodes of condomless receptive anal and vaginal sex with and without condoms; incidence of STI and HIV acquisition.

The investigators will employ a mixed ANOVA to look at intervention effects on adherence-as well as STI incidence, and safe sex practices-across time intervals. They will also estimate mixed regression models for the intervention.

ELIGIBILITY:
Inclusion Criteria

1. HIV- men and women, age 18 and higher, who are seeking PrEP and deemed appropriate per local site investigator following the CDC risk indication guidelines for PrEP.
2. Must fit into one of the study's CDC-identified risk strata: a) IDUs and/or b) Caucasian LGBTQ or Minority LGBTQ
3. Must be able to read and write English for themselves.

Exclusion Criteria

1. Same as that for PrEP initiation, e.g., existing HIV+ diagnosis or contra-indications, creatinine GFR < 60.
2. Current or previous use of PrEP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
PrEP Adherence | quarterly, for one year
  Tenofovir concentrations in dried blood spots

SECONDARY OUTCOMES:
HIV contraction | quarterly, for one year
  Diagnosis of HIV throughout the study period
Sexual Risk Behavior 1: Partners | quarterly, for one year
  Number of Partners in anal or vaginal sex
Sexual risk behavior 2: Condomless sex | quarterly, for one year
  number of condomless vaginal or anal sex occurrences
STI contraction | quarterly, for one year
  Diagnosis of an STI throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Nichole Ben Itzhak, PhD, Study Director — BI Development
Locations (1):
- Center for Inclusion Health, Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified information will be shared regarding STI/HIV diagnosis.